CLINICAL TRIAL: NCT06479252
Title: Comparing Centre-based, Remotely Supervised, and Self-administered Sit-to-stand Tests in Individuals With Chronic Respiratory Diseases
Brief Title: Comparing Centre-based, Remotely Supervised, and Self-administered STS Tests in Individuals With CRD
Acronym: STS24
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Dina Brooks, Senior Scientist, West Park Healthcare Centre, West Park Healthcare Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: WP-24-002
Record Dates: First submitted 2024-06-14; First posted 2024-06-28 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Chronic Lung Disease
Keywords: Assessment; Pulmonary Rehabilitation; Remote

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Centre-Based Condition (Active Comparator): Participants will be asked travel to West Park Healthcare Centre to complete the sit-to-stand (STS) tests under the supervision of a trained research team member. Participants will be guided through the standardized protocol for the STS tests.
  Interventions: Other: Sit-to-Stand Test (STS)
- Remotely Supervised Condition (Experimental): The sit-to-stand (STS) tests will be conducted in the patient's home and will be remotely monitored by a research staff member situated at the healthcare centre (via videoconference). The research team member will send a meeting invite to the participant who will independently join the videoconference from their home. At the onset of the study, participants will receive a handout to explain the materials they need to prepare for the session. Guidance will also be provided during the orientation meeting. Based on chair availability in participant's home, deviations will be noted by study staff. The testing procedure and instructions will be the same as the centre-based testing described.
  Interventions: Other: Sit-to-Stand Test (STS)
- Self-Administered Condition (Experimental): The self-administered sit-to-stand (STS) tests will be conducted independently by the patient in their home setting. No supervision will be provided by study staff during the testing sessions. At the onset of the study, participants will receive a handout to explain the materials they need to prepare for the session. Detailed instructions for completing the STS tests independently will be provided to the participant (Appendix B). Guidance will also be provided during the orientation meeting. The instructions and guide to self-administer the test will be piloted at the start of the study, and the content may be refined to meet the needs of patients.
  Interventions: Other: Sit-to-Stand Test (STS)

INTERVENTIONS:
Other: Sit-to-Stand Test (STS) — The 30-s and 1-min STS tests are reliable, valid, and responsive tests for measuring functional exercise capacity in patients with lung disease. For the STS tests that are centre-based or supervised remotely, investigators will collect the total number of repetitions on the 30-s and 1-min STS tests, as well as the number and duration of rests within and between tests.

SUMMARY:
Despite evidence on the psychometric properties of sit-to-stand (STS) tests in chronic respiratory disease (CRD) populations, most studies have been conducted face-to-face. Given the recent emphasis on virtual pulmonary rehabilitation (VPR), there is a need to identify reliable and valid exercise tests that can be delivered in home-based settings, either supervised remotely or self-administered by patients. A repeated-measures crossover design will be used to test the home-based administration of STS tests. The 30-second STS (30-s STS) and 1-minute STS (1-min STS) tests will be randomly administered across three test conditions (centre-based, remotely supervised, and self-administered). Data will summarize the feasibility of remotely supervised and self-administered STS tests and compare the performances of centre-based tests with remotely supervised and self-administered versions of STS tests in patients with CRD.

DETAILED DESCRIPTION:
This study aims to assess the implementation and measurement of both the 30s-STS and the 1-min STS tests when remotely supervised or self-administered in individuals with CRD. More specifically, the objectives of this study are as follows:

i. To explore the feasibility, acceptability, and implementation of remotely supervised and self-administered STS tests in individuals with CRD.

ii. To evaluate whether STS test performance differs by mode of administration (1: centre-based, 2: remotely supervised, and 3: self-administered) in individuals with CRD.

iii. To investigate the clinical utility of remotely supervised and self-administered STS tests as a measure of functional status among in individuals with CRD.

A repeated-measures crossover design will be used. The 30-s STS and the 1-min STS tests will be administered to participants across three test conditions (centre-based, remotely supervised, and self-administered).

At the onset of the study, participants will attend an initial orientation meeting over videoconference (approximately 30 minutes) to review the process of the study and data collection. The orientation meeting will include instruction on completing the STS tests at home, and participants will demonstrate a repetition of the STS. Prior to completing the STS testing, each participant will self-report their functional status using the modified version of the Pulmonary Functional Status and Dyspnea Questionnaire and demographic/descriptive measures will be collected from the participant's clinical record. Participants will complete the STS tests (30-second and 1-minute) across three conditions (centre-based, remote, self-administered). The test order will be randomized by condition and will be completed on separate days. For each testing condition, the 30-s STS and 1-min STS tests will be completed in random order. All tests will occur over a maximum 7-day period. Neither the study staff nor the participants will be blinded to the order of their tests. Blood oxygen level (SpO2), heart rate (HR) and level of dyspnea (Borg scale) will be recorded before and immediately after each test. On each test day, participants will be given a 5-min rest period between each STS test protocol. Before starting the second test, participants will indicate that they feel ready to start and study staff will confirm participants' oxygen level, HR and dyspnea have returned to pre-test levels. Delays in starting time past the 5-min rest period will be documented by research staff. After completing three testing conditions, participants will complete a questionnaire regarding feasibility and acceptability of different testing conditions.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of chronic respiratory disease (e.g., Chronic Obstructive Pulmonary Disease, Interstitial Lung Disease, Asthma).
* Male and female patients ≥18 years of age.
* Able to perform at least 5 repetitions in the 1-min sit-to-stand test without use of upper extremities.
* Access to a portable pulse oximeter at home to measure heart rate and oxygen saturation.
* Access to technology for remote supervision (e.g., mobile phone, laptop/computer, iPad)

Exclusion Criteria:

* Lower limb surgery in the preceding 3 months.
* Medically unstable to perform exercise tests (e.g., no exacerbation in the preceding two weeks).
* Predominant neurological or musculoskeletal limitations to completing sit-to-stand.
* At risk of falling during sit-to-stand due to impaired balance, as indicated in their clinical record, and/or PR assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
30 second Sit-to-Stand Test | Over a 7 day period, outcome will be collected at three time points (e.g., once within each testing condition: centre-based, remote, and self-administered)
  The 30-s and 1-min STS tests are reliable, valid, and responsive tests for measuring functional exercise capacity in patients with lung disease. For the STS tests that are centre-based or supervised remotely, investigators will collect the total number of repetitions on the 30-s and 1-min STS tests, as well as the number and duration of rests within and between tests. Scores on the STS tests will be recorded using the data collection form.
1 minute Sit-to-stand Test | Over a 7 day period, outcome will be collected at three time points (e.g., once within each testing condition: centre-based, remote, and self-administered)
  The 30-s and 1-min STS tests are reliable, valid, and responsive tests for measuring functional exercise capacity in patients with lung disease. For the STS tests that are centre-based or supervised remotely, investigators will collect the total number of repetitions on the 30-s and 1-min STS tests, as well as the number and duration of rests within and between tests. Scores on the STS tests will be recorded using the data collection form.

SECONDARY OUTCOMES:
Oxygen Saturation (Sp02) | participants will be asked to record their oxygen saturation (Sp02) before and after the STS test (30 second and 1 minute) within each arm
  Oxygen saturation (Sp02) will be measured using a finger pulse oximeter before and after the 30-s and 1-min STS. Self-monitoring using remote pulse oximetry has been shown to be feasible and accurate in CRD populations. The oximeter will provide a printout of values reflecting oxygen level, which will be transcribed to a data collection form. Patients will be asked to use their own pulse oximeter, and the make and model will be recorded by study staff.
Heart Rate | Participants will be asked to record their heart rate before and after the STS test (30 second and 1 minute) within each arm
  Heart rate will be measured using a finger pulse oximeter before and after the 30-s and 1-min STS tests. Self-monitoring using remote pulse oximetry has been shown to be feasible and accurate in chronic respiratory disease populations. The oximeter will provide a printout of values reflecting HR, which will be transcribed to a data collection form. Patients will be asked to use their own pulse oximeter, and the make and model will be recorded by study staff.
Modified Borg Scale | participants will be asked to record their data pre-and post STS test (30 second and 1 minute) within each arm
  The Modified Borg Dyspnea scale is a self-reported measure of one's difficulty breathing upon exertion. The instrument provides a standard method for patients to select ratings of dyspnea on a scale based on descriptors that correspond to specific numbers. At the start and at the end of each STS test, subjects will rate their perceived rate of dyspnea ("difficulty breathing") using the modified Borg Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Brooks, PhD, Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No